CLINICAL TRIAL: NCT02297880
Title: Effects of Beverages Containing Low Calorie Sweeteners (LCS) on Energy and Macronutrient Intakes and on Hunger, Appetite and Satiety Sensations
Brief Title: Effects of Low Calorie Sweeteners on Dietary Intakes, Hunger, Appetite and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Coca-Cola Company (Industry)
Collaborators: CreaBIO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CreaBIO1
Record Dates: First submitted 2014-11-13; First posted 2014-11-21 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Eating Behavior
Keywords: low calorie sweetener satiety, intake, hunger
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beverage containing low calorie sweeteners (Experimental): Beverage containing low calorie sweeteners (flavour)
  Interventions: Other: Beverage containing low calorie sweeteners
- Still water (Active Comparator): Still water (no flavour)
  Interventions: Other: Still water

INTERVENTIONS:
Other: Beverage containing low calorie sweeteners — Beverage containing low calorie sweeteners
  Arms: Beverage containing low calorie sweeteners
Other: Still water — Still water (no flavour)
  Arms: Still water

SUMMARY:
Although there is evidence that low calorie sweeteners (LCS) do not stimulate hunger or appetite, divergent opinions appear regularly both in the scientific literature and in the popular press. The goal of this study is to examine the effects of LCS containing beverages on appetite and intake in healthy individuals.

DETAILED DESCRIPTION:
The study will be a monocentric randomized controlled open trial including two parallel groups to examine effects of LCS beverages as compared to water on daily intakes of energy and macronutrients. The effects of LCS beverages on hunger, satiety, desire to eat and on the selection of sweet or savory foods eating occasions will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index: Lower limit 18 kg/m²; Upper limit 28 kg/m²; weight stable within ± 3 kg in the last 6 months
* Habitual energy intake within the 95% confident interval of the reference energy intake for the French population (as provided by the INCA 2 survey
* Must not be a regular drinker of LCS beverages (less than once a week no more than every 15 days) and be willing to use LCS according to protocol
* For female participants: not pregnant, not breast feeding, planning to become pregnant during the study or on contraception since at least 3 months (regular 28-day cycle)
* Subject registered with the French Social Security.

Exclusion Criteria:

* Currently diagnosed somatic pathology
* On medication affecting metabolism, weight, energy intake, or energy expenditure in the last 6 months
* Major psychiatric disorder, particularly eating disorders as defined by the Diagnostic and Statistical Manual od Mental Disorders-IV
* Rejection of sweet foods or drinks as revealed by the diet history
* Smoking subject planning to stop smoking in the next 3 months
* Subjects suffering from food allergies or intolerance
* Subject not capable of understanding the constraints of the study and who not agree to abide

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Subjective sensations: hunger, satiety and desire to eat | 9 weeks
  Visual Analog Scales

SECONDARY OUTCOMES:
Energy and macronutrient intakes | 9 weeks
  Diet history questionnaire
Anthropometric parameters | 9 weeks
  body weight, height, waist and hip circumferences

CONTACTS AND LOCATIONS:
Locations (1):
- CreaBio Rhône-Alpes laboratory, 9 avenue du Professeur Fleming, Givors, Lyon, France

REFERENCES:
- [Derived] Fantino M, Fantino A, Matray M, Mistretta F. Beverages containing low energy sweeteners do not differ from water in their effects on appetite, energy intake and food choices in healthy, non-obese French adults. Appetite. 2018 Jun 1;125:557-565. doi: 10.1016/j.appet.2018.03.007. Epub 2018 Mar 9. PMID 29526693